CLINICAL TRIAL: NCT02984852
Title: A Single-dose, Open-label, Randomized, Crossover Study to Assess the Relative Bioavailability of the Fixed-dose Combination Tablet Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Administered Orally as a Whole Tablet, as a Split Tablet, and as Crushed Tablet in Healthy Subjects
Brief Title: Study to Evaluate the Relative Bioavailability of Fixed-dose Combination Tablet Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) as a Whole Tablet, as a Split Tablet, and as Crushed Tablet in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108258; TMC114FD2HTX1004 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Darunavir; Cobicistat; Emtricitabine; Racivir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (6):
- Treatment sequence ABC (Experimental): Participants will receive a single oral tablet of darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF fixed dose combination [FDC]) Treatment A (whole tablet) as reference in session 1 then Treatment B(split tablet) as test in session 2 followed by Treatment C (crushed tablet mixed in applesauce) as test in session 3 under fed conditions (standardized breakfast) on Day 1 of each treatment session. There will be a washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)
- Treatment sequence ACB (Experimental): Participants will receive a single oral tablet of D/C/F/TAF [FDC] Treatment A in treatment session 1, then Treatment C in session 2 followed by Treatment B in session 3 under fed conditions (standardized breakfast) on Day 1 with washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)
- Treatment sequence BCA (Experimental): Participants will receive a single oral tablet of D/C/F/TAF [FDC] Treatment B in session 1 then Treatment C in session 2 followed by Treatment A in session 3 under fed conditions (standardized breakfast) on Day 1 with washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)
- Treatment sequence BAC (Experimental): Participants will receive a single oral tablet of D/C/F/TAF [FDC] Treatment B in session 1 then Treatment A in session 2 followed by Treatment C in session 3 under fed conditions (standardized breakfast) on Day 1 with washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)
- Treatment sequence CAB (Experimental): Participants will receive a single oral tablet of D/C/F/TAF [FDC] Treatment C in session 1 then Treatment A in session 2 followed by Treatment B in session 3 under fed conditions (standardized breakfast) on Day 1 with washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)
- Treatment sequence CBA (Experimental): Participants will receive a single oral tablet of D/C/F/TAF [FDC] Treatment C in session 1 then Treatment B in session 2 followed by Treatment A in session 3 under fed conditions (standardized breakfast) on Day 1 with washout period of at least 7 days between consecutive drug intakes.
  Interventions: Drug: Darunavir (DRV); Drug: Cobicistat (COBI); Drug: Emtricitabine (FTC); Drug: Tenofovir Alafenamide (TAF)

INTERVENTIONS:
Drug: Darunavir (DRV) — Darunavir 800 milligram (mg) will be taken orally in FDC together with COBI(150mg)/FTC(200mg)/TAF(10mg).
Drug: Cobicistat (COBI) — Cobicistat 150 milligram (mg) will be taken orally in FDC together with DRV(800mg)/FTC(200mg)/TAF(10mg).
Drug: Emtricitabine (FTC) — Emtricitabine 200 milligram (mg) will be taken orally in FDC together with COBI(150mg)/DRV(800mg)/TAF(10mg).
Drug: Tenofovir Alafenamide (TAF) — Tenofovir Alafenamide 10 milligram (mg) will be taken orally in FDC together with COBI(150mg)/FTC(200mg)/DRV(800mg).

SUMMARY:
The purpose of this study is to evaluate the single-dose pharmacokinetics and relative bioavailability of Darunavir (DRV) 800 milligram (mg), Cobicistat (COBI) 150 mg, Emtricitabine (FTC) 200 mg, and tenofovir alafenamide (TAF) 10 mg when administered as a fixed-dose combination (FDC) (D/C/F/TAF) tablet in healthy adult participants when given as Treatment A (reference): a single dose of D/C/F/TAF (800/150/200/10 mg) FDC tablet swallowed as a whole, intact tablet with 240milliliter (mL) of noncarbonated water.Treatment B (test): a single dose of D/C/F/TAF (800/150/200/10 mg) FDC tablet as a split tablet swallowed with 240 mL of noncarbonated water. Treatment C (test): a single dose of D/C/F/TAF (800/150/200/10 mg) FDC tablet as a crushed tablet mixed in 4 ounces (oz) of applesauce.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months prior to selection
* Body mass index (BMI) of 18.0 to 32 kilogram per square meter (kg/m^2), inclusive
* Woman must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening and a negative sensitive urine pregnancy test on Day -1 before the first dose of study drug
* Woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, a non-vasectomized man who is sexually active with a woman of childbearing potential must agree to use a highly effective barrier method of contraception

Exclusion Criteria:

* Positive human immunodeficiency virus -1 (HIV-1) or HIV-2 test at screening
* Hepatitis A, B, or C infection, confirmed by a positive hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) test, respectively, at screening
* History of renal insufficiency
* History of significant drug-induced skin reactions (such as, but not limited, to Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), and/or erythema multiforme) or history of allergies to drugs (such as, but not limited to, sulfonamides and penicillins)
* Previously participated in a multiple-dose study with Darunavir (DRV), Cobicistat (COBI), Emtricitabine (FTC), Tenofovir Alafenamide (TAF), or Tenofovir Disoproxil Fumarate (TDF)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 4
  Cmax is defined as the maximum observed plasma concentration.
Area Under the Plasma Concentration Curve from time zero to the last quantifiable (AUC [0-last]) | Up to Day 4
  AUC (0-last) is the area under the Plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 4
  The AUC (0-infinity) is the area under the plasma concentration time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Screening (21 days ) to End of the study (7 to 10 days after the last dose)
Number of Participants With Clinical Laboratory Results as a Measure of Safety and Tolerability | Screening (21 days ) to End of the study (7 to 10 days after the last dose)
Number of Participants With Vital Signs as a Measure of Safety and Tolerability | Screening (21 days ) to End of the study (7 to 10 days after the last dose)
Number of Participants With Physical Examination Findings as a Measure of Safety and Tolerability | Screening (21 days ) to End of the study (7 to 10 days after the last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Tempe, Arizona, United States